CLINICAL TRIAL: NCT03885141
Title: Phase II / III Study, One Center, Double-Blind, With Placebo Use, in Parallel Groups to Assess the Efficacy and Safety of Zolpidem® Orodispersible in Adult Subjects (Females and Males) in the Treatment of Maintenance Insomnia Disorder.
Brief Title: Biolab Zolpidem Orodispersible 1.0 mg, 1.75 mg and 3.5 mg to Treat Maintenance Insomnia Disorder.
Acronym: ZOLP_18_01
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Biolab Sanus Farmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZOLP_18_01
Record Dates: First submitted 2019-03-14; First posted 2019-03-21 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Insomnia Disorder
Keywords: Insomnia; Zolpidem
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Zolpidem

STUDY DESIGN:
Intervention Model Description: Assessment of the efficacy of Zolpidem treatment. The following will be evaluated: improvement of maintenance insomnia through the Sleep Diary and the Severity Index of the Insomnia (IGI), as well as sleep latency through polysomnography and treatment safety through the reporting of adverse events and laboratory tests.
Who Masked: Participant, Investigator
Masking Description: Placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Men - Placebo (Placebo Comparator): Men - Placebo, 1 tablet if a wake up occurs
  Interventions: Drug: Zolpidem
- Men - Zolpidem 1.75 mg (Experimental): Men - Zolpidem 1.75 mg, 1 tablet if a wake up occurs
  Interventions: Drug: Zolpidem
- Men - Zolpidem 3.5 mg (Experimental): Men - Zolpidem 3.5 mg, 1 tablet if a wake up occurs
  Interventions: Drug: Zolpidem
- Women - Placebo (Placebo Comparator): Women - Placebo, 1 tablet if a wake up occurs
  Interventions: Drug: Zolpidem
- Women - Zolpidem 1.0 mg (Experimental): Women - Zolpidem 1.0 mg, 1 tablet if a wake up occurs
  Interventions: Drug: Zolpidem
- Women - Zolpidem 1.75 mg (Experimental): Women - Zolpidem 1.75 mg, 1 tablet if a wake up occurs
  Interventions: Drug: Zolpidem

INTERVENTIONS:
Drug: Zolpidem — Zolpidem or Placebo if there is a wake up during the night

SUMMARY:
Biolab Sanus is developing a product in the form of orodispersible tablet containing 1.0 mg, 1.75 mg and 3.5 mg of Zolpidem®. Thus, it is intended to evaluate the efficacy of Zolpidem® Orodispersible 1.0 mg or 1.75 mg in women and Zolpidem Orodispersible 1.75 mg or 3.5 mg in men for the improvement of the maintenance insomnia disorder, through the evaluation of the Insomnia Severity Index, and using a Sleep Diary throughout the study, as well as to evaluate the latency of the sleep after a spontaneous or provoked wake up measured by polysomnography.

DETAILED DESCRIPTION:
Information provided evidence for the therapeutic use of Zolpidem® in the treatment of insomnia. Several studies have emphasized the importance of using Zolpidem® in small doses, in the orodispersible form, in the treatment of insomnia. Accordingly, Biolab Sanus is developing a product in the form of orodispersible tablet containing 1.0 mg, 1.75 mg and 3.5 mg of Zolpidem®. Thus, it is intended to evaluate the efficacy of Zolpidem® Orodispersible 1.0 mg or 1.75 mg in women and Zolpidem Orodispersible 1.75 mg or 3.5 mg in men for the improvement of the maintenance insomnia disorder, through the evaluation of the Insomnia Severity Index, and using a Sleep Diary throughout the study, as well as to evaluate the latency of the sleep after a spontaneous or provoked wake up measured by polysomnography.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 18 years and ≤ 64 years of age
2. Participants willing and able to provide a written informed consent form, after an explanation of the nature of the study, and prior to any procedures related to the study.
3. Adults with clinical diagnosis of insomnia, as defined by the Diagnostic and Statistical Manual of Mental Disorders (DSM-V-TR) and who complain of difficulty in maintaining sleep, starting more than three months before the study initiation, and for three or more sleepless nights per week.
4. Participants with ability to understand and willingness to comply with the study procedures

Exclusion Criteria:

1. History of Allergy or Hypersensitivity to Zolpidem;
2. All initial and secondary insomnia;
3. Basal polysomnography with apnea and hypopnea index> 20 events / hour and PLM (Periodic Leg Movements)> 15 events / hour.
4. Participants who used central nervous system medication or other medication known to interfere with the sleep / wake up cycle within 15 days prior to enrollment in the study, at the discretion of the study investigator.
5. Clinically significant diseases or surgeries, at the discretion of the principal investigator, within 30 days prior to study inclusion.
6. History of chemical dependence or alcohol abuse.
7. Any significant neurological and psychiatric disease or laboratory findings present, unless adequately controlled with medication allowed in the protocol.
8. Participants who received any investigational medication in the last 12 months prior to study inclusion.
9. Women who are pregnant or breastfeeding or who wish to become pregnant or who refuse to use safe contraceptive methods during the study.
10. Any disorder of the circadian cycle.
11. Regular night shift work within the last 2 weeks prior to study enrollment or expected to work in shifts during the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Men: Placebo or Zolpidem 1.75 mg or Zolpidem 3.5 mg
  Women: Placebo or Zolpidem 1.0 mg or Zolpidem 1.75 mg
Enrollment: 366 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Difference Insomnia Severity Index (ISI) as assessed by questionnaire before treatment and after the treatment | 28 days
  To analyse the efficacy of Zolpidem® Orodispersible treatment 1.0 mg or 1.75 mg in women and 1.75 mg and 3.5 mg in men, compared to placebo, after taking the medication when a spontaneous wake up occurs during 28 days. The assessement will be performed by means of the standard questionnaire before and at the end of the treatment period. The computed mean difference for each treatment will be compared by ANOVA (treatment doses vs placebo in each gender) in order to assess its statistical significance.

SECONDARY OUTCOMES:
Total Sleep Time (polysomnography parameter) | 1 day
  Total Sleep Time after a provoked wake up, and the administration of 1 tablet of Zolpidem® Orodispersible 1.0 mg or 1.75 mg in women and 1.75 mg or 3.5 mg in men, as compared to placebo administration after a provoked wake up.
Sleep Efficiency (polysomnography parameter) | 1 day
  Sleep Efficiency after a provoked wake up, and the administration of 1 tablet of Zolpidem® Orodispersible 1.0 mg or 1.75 mg in women and 1.75 mg or 3.5 mg in men, as compared to placebo administration after a provoked wake up.
Sleep Latency (polysomnography parameter) | 1 day
  Sleep Latency after a provoked wake up, and the administration of 1 tablet of Zolpidem® Orodispersible 1.0 mg or 1.75 mg in women and 1.75 mg or 3.5 mg in men, as compared to placebo administration after a provoked wake up.

IPD SHARING:
Plan to Share IPD: No